CLINICAL TRIAL: NCT04624126
Title: Non-invasive External Device for Erectile Dysfunction (3D-Erect): a Pilot Study
Brief Title: External Device for Erectile Dysfunction (3D-Erect)
Acronym: 3D-Erect
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Michael Eisenberg, Associate Professor of Urology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB-57222
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Erectile Dysfunction; Impotentia Erigendi
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- 3D-Erect arm (Experimental): Participants will be asked to use the 3D-printed penile device during their intercourse with partners.
  Interventions: Device: 3D-Erect

INTERVENTIONS:
Device: 3D-Erect — 3D-printed erectile device for intercourse

SUMMARY:
The aim of this clinical trial is to test the safety and feasibility of a non-invasive 3D-printed external penile device to achieve successful and satisfactory sexual intercourse in men with erectile dysfunction (ED).

DETAILED DESCRIPTION:
A clinical trial to test the safety and feasibility of our newly developed non-invasive 3D-printed external penile device for the treatment and recovery of erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* males >18 years old suffering from any cause moderate to severe erectile dysfunction (e.g. ED after radical prostatectomy and/or radiation therapy for prostate cancer and or other pelvic malignancies affecting the sexual potency; emotional and psychological ED; organic vascular and/or metabolic ED etc.)
* having a female partner willing to participate in the study.

Exclusion Criteria:

* not willing to attempt sexual vaginal intercourse with their partner
* inability to wear/operate the external penile device for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in modified International Index of Erectile Dysfunction score | baseline and up to 1 month post-baseline
  score 0 to 30 with higher score meaning overall better erectile function

CONTACTS AND LOCATIONS:
Overall Officials: Michael Eisenberg, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care, Stanford Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No